CLINICAL TRIAL: NCT05668884
Title: Effects and Safety of GEMOX Combined With Donafenib and Tislelizumab in Advanced Biliary Tract Carcinoma：a Prospective, Single-arm, Multi-center Phase II Study
Brief Title: GEMOX Combined With Donafenib and Tislelizumab in Advanced Biliary Tract Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2209260-22-2407A
Record Dates: First submitted 2022-12-12; First posted 2022-12-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Biliary Tract Carcinoma
Keywords: Donafenib; Tislelizumab; Effects; Safety
MeSH Terms: interventions — Oxaliplatin; donafenib; tislelizumab

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Combination of Gemox, Donafenib and Tislelizumab
  Interventions: Combination Product: Combination of Gemcitabine, Oxaliplatin, Donafenib and Tislelizumab

INTERVENTIONS:
Combination Product: Combination of Gemcitabine, Oxaliplatin, Donafenib and Tislelizumab — Combination of Gemcitabine, Oxaliplatin, Donafenib and Tislelizumab every 3 weeks

SUMMARY:
In this phase 2 study, the investigators aim to evaluate the effects and safety of combined therapy using oxaliplatin and gemcitabine chemotherapy, Donafenib and Tislelizumab for patients with advanced biliary tract carcinoma.

DETAILED DESCRIPTION:
Most advanced biliary tract carcinoma (BTC) patients are often accompanied by local or distant metastases and lose the opportunity for surgical resection. For patients with advanced BTC who have been in stages III and IV (AJCC/UICC, V2, 2018), the survival time is less than 4 months, and there is currently no standard treatment. The Gemox chemotherapy (oxaliplatin + gemcitabine) has been used in the treatment of advanced BTC, but the efficacy is still unsatisfactory. Donafenib is a small molecule multi-kinase inhibitor, the main targets including VEGFR1-3, PDGFRα, RET(ret proto-oncogene ), c-KIT(KIT proto-oncogene, receptor tyrosine kinase), Raf,FLT3,have anti-angiogenic effects, have been proven effective in hepatocellular carcinoma. In recent years, monoclonal antibodies against programmed cell death protein 1 (PD1) have shown remarkable therapeutic effects in the treatment of various solid tumors. Prior to this, the combined treatment of GEMOX combined with Donafenib and Tislelizumab was proved satisfying safety. Meanwhile,the phase-I trial showed good efficacy in conversion rate and 6-month overall survival rate. Due to the limitted small sample size of the phase I trial, the investigators aim to expand the sample size to further verify the effects and safety of combined therapy in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤75 years;
* ECOG physical condition score: 0~1;
* Histologically or cytologically confirmed advanced biliary tract carcinoma (including gallbladder, intrahepatic and extrahepatic cholangiocarcinoma);
* Preoperative imaging assessment of the disease stage was III/IV;
* At least one measurable lesion (according to mRECIST criteria)
* Child-Pugh classification : A or B
* The main organs function well, and the examination indicators meet the following requirements:
* Routine blood tests: Hemoglobin ≥90 g/L (no blood transfusion within 14 days);Neutrophil count ≥1.5×10^9/L; Platelet count ≥80×10^9/L;
* Biochemical examination: Total bilirubin ≤2×ULN (upper normal value); ALT or AST ≤ 2.5×ULN; Endogenous creatinine clearance ≥ 50 mL /min (Cockcroft-Gault formula);
* thyroid function:Thyroid function is normal, thyroid stimulating hormone TSH is defined to be within the normal range. If baseline TSH is outside the normal range, T3 and T4 can be included if they are within the normal range;
* Myocardial enzyme profile:The myocardial enzyme profile was in the normal range (if simple laboratory abnormalities that were not clinically significant as determined by the investigators could also be included);
* Estimated survival time ≥ 3 months;
* Sign the informed consent voluntarily;
* Good compliance, and family members willing to cooperate with follow-up.

Exclusion Criteria:

* Patients with other uncured malignant tumors;
* Pregnant or lactating women who are required to withdraw from the clinical trial if they become pregnant during the study period;
* Previous antitumor therapy for the disease in this study;
* Participated in clinical trials of other drugs within one month;
* Patients with a known history of other systemic serious diseases before screening;
* Obstructive jaundice (after active treatment such as biliary drainage or stent, the patients can be included in the group after the liver function returns to normal);
* Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number greater than the upper limit of normal in the clinical laboratory of the study center);
* Active HCV infected persons (HCV antibody positive with HCV RNA levels above the lower limit of detection);
* Allergic to any investigational drug or excipient;
* Long-term unhealed wounds or incomplete healing fractures;
* Previous organ transplantation history;
* Having a history of abuse of psychotropic substances and being unable to quit or having mental disorders;
* A history of immune deficiency or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* Concomitant conditions that, in the investigator's judgment, seriously endanger the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 6 months
  objective response rate(ORR)，defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1

SECONDARY OUTCOMES:
1-year Recurrence free survival | 1 year
  1-year Recurrence free survival
Progression-free survival | 6 months
  progression-free survival(PFS), defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
Overall survival | 6 months
  overall survival(OS), defined as the time from enrollment to death due to any cause.
Incidence and degree of Adverse Events and Serious Adverse Events | 6 months
  Incidence, severity, and relationship to study drugs of all adverse events (AEs), treatment-related adverse events (TRAEs), and serious adverse events (SAEs).
Conversion rate | 6 months
  Conversion rate, defined as the percentage of the conversion of patients with BTC assessed as unresectable into resectable through interventions, including the conversion of unresectable into resectable in the scientific sense such as insufficient future liver remnant(FLR), as well as the conversion of R1 and R2 to R0.

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Zhao, M.D., Study Director — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No